CLINICAL TRIAL: NCT00810394
Title: Single Agent Sorafenib in Advanced Solid Tumors: Phase II Evaluation of Dose Re-Escalation Following a Dose Reduction (IST000375)
Brief Title: Sorafenib in Treating Patients With Advanced Malignant Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#213; 236614 (Other: University of California Davis); IST000375 (Other Grant/Funding Number: Bayer); UCDCC-213 (Other: University of California Davis)
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2017-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sorafenib (Experimental): Dose Re-Escalation Following a Dose Reduction
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Patients will be registered and started on the standard recommended dose-schedule for sorafenib (400 mg tablet by mouth twice a day continuously). Dose reductions will be instituted in the event of grade 3 or higher hematologic or non-hematologic toxicity or for any toxicity that is considered by the patient or physician as intolerable.
  Other Names: Nexavar

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying the side effects and best dose of sorafenib and to see how well it works in treating patients with advanced malignant solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the feasibility of re-escalating the dose of sorafenib tosylate in patients with advanced malignant solid tumors who initially required a dose reduction for toxicity, and dose escalation in those patients who are able to tolerate the initial dose.

Secondary

* To evaluate the efficacy of this drug in these patients who are able to tolerate a dose escalation initially or after a dose reduction compared to those who are unable to tolerate a dose escalation.

Tertiary

* To evaluate the percentage and demographic characteristics of patients who are able to tolerate 2 dose escalations without a dose reduction.

OUTLINE: This is a dose-finding study.

* Course 1: Patients receive oral sorafenib tosylate twice daily at dose level 0 on weeks 1-4.
* Course 2: Patients experiencing no dose-limiting or intolerable toxicities receive oral sorafenib tosylate at dose level +1 twice daily on weeks 5-8; while patients experiencing dose-limiting or intolerable toxicities receive oral sorafenib tosylate at dose level -1 once daily on weeks 5-8.
* Course 3: Depending on whether or not patients are experiencing dose-limiting or intolerable toxicities, they are escalated to dose level 0 or dose level +2 (patients in both dose levels receive oral sorafenib tosylate twice daily) in weeks 9-12, or de-escalated to dose level 0 or dose level -2 (patients in dose level -2 receives oral sorafenib tosylate once every other day) in weeks 9-12.
* Maintenance therapy: Patients receive oral sorafenib tosylate at the dose level* attained at the end of course 3. Treatment continues in the absence of unacceptable toxicity.
* Dose level de-escalation for toxicity or dose re-escalation after a toxicity-related dose reduction allowed to a maximum level of the initial dose level of the maintenance therapy.

After completion of study therapy, patients are followed for up to 1 year.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed metastatic or unresectable solid tumor for which standard curative or palliative measures do not exist or are no longer effective or solid tumor for which sorafenib is considered acceptable therapy
* Age > 18 years old
* Performance Status 0 - 2
* Measurable or non-measurable disease.
* Adequate bone marrow, liver and renal function
* Any number of prior chemotherapy regimens are allowed.
* Any prior chemotherapy, immunotherapy or targeted therapy must have been completed at least 2 weeks prior to start of this protocol and all side effects resolved to grade 1 or less. Any prior radiation must have been completed at least 2 weeks prior to start of therapy.
* Women of childbearing potential must have a negative pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation. Men should use adequate birth control for at least three months after the last administration of sorafenib.
* Ability to understand and the willingness to sign a written informed consent.
* International normalized ratio < 1.5 or a Prothrombin Time/Partial thromboplastin time within normal limits.

Exclusion Criteria

* Prior therapy with sorafenib or sunitinib.
* Cardiac disease: Congestive heart failure > class II New York Heart Association.
* Symptomatic or uncontrolled brain metastasis.
* No component of squamous carcinoma can be present in any patient with non-small cell lung cancer
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Known HIV infection or chronic Hepatitis B or C.
* Active clinically serious infection > CTCAE Grade 2.
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding diathesis or coagulopathy
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first dose of study drug.
* Use of St. John's Wort or rifampin
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.
* Any condition that impairs patient's ability to swallow whole pills.
* Any significant malabsorption problem.
* Therapy with bevacizumab < 3 months prior to first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-12; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Primo N. Lara, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States

REFERENCES:
- [Result] Semrad TJ, Eddings C, Pan CX, Lau DH, Gandara D, Beckett L, Lara PN Jr. Feasibility study of intra-patient sorafenib dose-escalation or re-escalation in patients with previously treated advanced solid tumors. Invest New Drugs. 2012 Oct;30(5):2001-7. doi: 10.1007/s10637-011-9761-y. Epub 2011 Oct 21. PMID 22015991

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sorafenib
Started | 50
Cycle 2 600mg Twice Daily | 13
Cycle 2 400mg Once Daily | 22
Cycle 3 800 mg Twice Daily | 4
Cycle 3 400mg Twice Daily | 5
Completed | 47
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: With a sample size of 51 patients, this study has 90% power with an alpha of 0.05 to detect a dose re-escalation/escalation rate difference of 50% vs. 70%. If 31 or more patients are able to re-escalate successfully, the approach will be considered for further study.
Arm/Group | Sorafenib
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 61 [25 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Tolerating Re-escalated Dose of Sorafenib for 28 Days Without Dose Interruption or De-escalation for Toxicity
Description: Overall percentage of patients tolerating a dose escalation to 600 mg twice daily for 28 days plus the percentage tolerating a re-escalation to 400 mg twice daily in Cycle 3.
Time Frame: At least 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib
Number analyzed (Participants) | 50
Participants | 11

2. Secondary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR).
Time Frame: At least 3 months
Population: Of the 34 patients who were evaluable for treatment response by RECIST, no responses were observed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib
Number analyzed (Participants) | 34
Participants | 0

3. Secondary Outcome: Time to Disease Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib
Number analyzed (Participants) | 34
months | 4.7 [4.3 to 6.1]

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Sorafenib
Serious Adverse Events (participants affected / at risk) | 19/50
Other Adverse Events (participants affected / at risk) | 42/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=50)
Bronchopulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Fever (General disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1
Ataxia (Musculoskeletal and connective tissue disorders) | 1
INR (Blood and lymphatic system disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2
Skin Reaction (Skin and subcutaneous tissue disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Hand and Foot Syndrome (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=50)
Hemoglobin (Blood and lymphatic system disorders) | 10
Leukopenia (Blood and lymphatic system disorders) | 7
Lymphopenia (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Hypertension (Cardiac disorders) | 13
Fever (General disorders) | 5
Fatigue (General disorders) | 17
Weight Loss (General disorders) | 7
Dry Skin (Skin and subcutaneous tissue disorders) | 5
Hand Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 16
Pruritis (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 14
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Edema (Blood and lymphatic system disorders) | 3
Hypoalbuminemia (Blood and lymphatic system disorders) | 4
Alkaline Phosphatase (Blood and lymphatic system disorders) | 7
AST (Blood and lymphatic system disorders) | 5
Bicarbonate, Serum (Blood and lymphatic system disorders) | 4
Hyperbilirubinemia (Blood and lymphatic system disorders) | 3
Hyperkalemia (Blood and lymphatic system disorders) | 3
Hypokalemia (Blood and lymphatic system disorders) | 7
Hyponatremia (Blood and lymphatic system disorders) | 5
Hypophosphatemia (Blood and lymphatic system disorders) | 9
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2
Mood Alteration (Psychiatric disorders) | 4
Pain (General disorders) | 18
Voice Changes (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes